CLINICAL TRIAL: NCT05825638
Title: Evolution of Pulsed Oxygen Saturation Throughout an Interval Training Session Compared to a Continuous Training Session in Patients With Chronic Obstructive Pulmonary Disease With Exercise-induced Oxygen Desaturation.
Brief Title: Evolution of Pulsed Oxygen Saturation During Interval Training Compared to Continuous Training in COPD Patients
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier du Havre (Other)
Collaborators: Medrinal Clement (Unknown); Combret Yann (Unknown); Machefert Margaux (Unknown)
Responsible Party: Principal Investigator, Guillaume Prieur, Principal Investigator, Groupe Hospitalier du Havre
Other Study IDs: 2022-A02087-36
Record Dates: First submitted 2023-01-10; First posted 2023-04-24 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: COPD; Exercise; Pulmonary Rehabilitation; Desaturation of Blood
Keywords: COPD; Pulmonary rehabilitation; Interval training
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Continuous training session
  Interventions: Other: Continuous training session
- Interval Training session
  Interventions: Other: Interval training session

INTERVENTIONS:
Other: Continuous training session — Continuous training consists of a 5 minute warm up, 5 minute cool down and 20 minutes of moderate intensity work. The workload is set at 60% of the patient's maximum power
  Groups: Continuous training session
Other: Interval training session — Interval training consists of a 5-minute warm-up, a 5-minute cool-down and 20 minutes of alternating 60 seconds of high-intensity work (100% of the maximum power recorded in the incremental test that was carried out when the patient was admitted to the pulmonary rehabilitation department) and 60 seconds of unloaded pedalling or rest.
  Groups: Interval Training session

SUMMARY:
A problem often observed during exercise training is oxygen desaturation exclusively during exercise in some patients. In the case of exercise-induced desaturation, it may be suggested to train these patients in interval training to limit exercise-induced desaturation. Interval training consists of alternating active phases of short duration (often 30 seconds to 1 minute) followed by a short active or passive recovery phase of equivalent duration to the previous phase. Investigators therefore hypothesise that interval training on a cycloergometer or treadmill can limit exercise-induced desaturation in COPD patients.

The aim of the study is to observe the evolution of pulsed oxygen saturation between a continuous training session and a interval training session.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of COPD
* participating in a pulmonary rehabilitation programme
* with an exercise-induced desaturation less than 90%
* no oxygen supplementation

Exclusion Criteria:

* Under 18 years of age
* Pregnant woman
* Person not affiliated to a health insurance regime or not benefiting from a social security regime
* Patient under curatorship, guardianship or safeguard of justice
* Patient speaking a language other than French
* Patient with severe hypoxaemia (SpO2 ≤ 80%) during exercise
* Patient having had a moderate or severe exacerbation (hospitalisation for respiratory reasons) in the previous 4 weeks
* Patients with orthopaedic, rheumatic, vascular or neurological pathology limiting their ability to make an effort
* Breastfeeding women

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with COPD who meet the inclusion criteria will be offered to participate in this study during a pulmonary rehabilitation programme which will take place in the pneumology rehabilitation department of the Le Havre Hospital. If the patient wishes to participate in the study, he/she will be given an information note containing a declaration of non-opposition which he/she will have to complete and sign.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-10-10 (Actual)

PRIMARY OUTCOMES:
Difference in oxygen pulsed saturation | One week
  Difference in minimum saturation during both exercise, the measurement will be performed with a pulse oximeter (Spirodoc, MIR)

SECONDARY OUTCOMES:
Difference in oxygen pulsed saturation | One week
  Difference in mean pulsed oxygen saturation and the time spent with a pulsed oxygen saturation below 90% during the two training sessions. The measurement will be performed with a pulse oximeter (Spirodoc, MIR)
Difference in peripheral muscle oxygenation | One week
  Muscle oxygenation (arbitrary unit) will be evaluated using Near-infrared spectroscopy technology. the measurement will be performed with a Near Infrared spectroscopy (Portamon, Artinis Medical Systems)
Difference in respiratory rate | One week
  Difference in respiratory rate will be measured breath-by-breath using a portable spirometer (Spirodoc, MIR)
Difference in tidal volume | One week
  Difference in tidal volume will be measured breath-by-breath using a portable spirometer (Spirodoc, MIR)
Difference in inspiratory capacity | One week
  Difference in inspiratory capacity will be measured using a portable spirometer (Spirodoc, MIR)
Difference in Dyspnea | One week
  Dyspnea peak during exercise using the modified Borg scale 0-10, 0 no dyspnea, 10 maximal dyspnea
Difference in muscle discomfort | One week
  Muscle discomfort peak during exercise using the modified Borg scale 0-10, 0 no dyspnea, 10 maximal dyspnea

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Prieur, PT, PhD, Principal Investigator — Groupe Hospitalier du Havre
Locations (1):
- Groupe Hospitalier du Havre, Le Havre, Normandy, France

IPD SHARING:
Plan to Share IPD: Yes
deidentified participtant data
Supporting Information: SAP, CSR
Time Frame: after publication
Access Criteria: the request shall be sent to Guillaume Prieur (gprieur.kine@gmail.com)